CLINICAL TRIAL: NCT04191577
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of CVN424 in Parkinson's Disease Patients With Motor Fluctuations
Brief Title: Study of CVN424 in Parkinson's Disease Patients With Motor Fluctuations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cerevance Beta, Inc. (Industry)
Responsible Party: Sponsor
Organization: Cerevance (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVN424-201
Record Dates: First submitted 2019-10-30; First posted 2019-12-10 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Planned dose levels are placebo, low dose, and high dose of CVN424. Study drug dispensed as CVN424 suspension (or matching placebo) in amber glass bottles suitable for self-administered dosing.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo to be administered once daily.
  Interventions: Drug: Placebo
- CVN424 (Low Dose) (Active Comparator): Low dose of CVN424 to be administered once daily.
  Interventions: Drug: CVN424 Low Dose
- CVN424 (High Dose) (Active Comparator): Patients randomized to the high dose will receive low-dose CVN424 once daily from day 1 to day 7, and will then increase their dose to the full high-dose once daily beginning on day 8.
  Interventions: Drug: CVN424 High Dose

INTERVENTIONS:
Drug: CVN424 Low Dose — CVN424
  Other Names: CVN424
  Arms: CVN424 (Low Dose)
Drug: CVN424 High Dose — CVN424
  Other Names: CVN424
  Arms: CVN424 (High Dose)
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a phase 2 study, randomized, double-blind, placebo-controlled, multicenter study of oral CVN424 at two dose levels (low-dose and high-dose) in Parkinson's disease (PD) patients with motor fluctuations.

DETAILED DESCRIPTION:
Approximately 135 male and female subjects with Parkinson's disease, on a stable dosage of levodopa but with an average of ≥ 2 h total OFF time/day and not less than 1 h per day, will be enrolled. Following baseline safety and efficacy assessments, subjects will be randomized to receive once-daily doses of either low-dose CVN424, high-dose CVN424, or matching placebo. All subjects not randomized to placebo will initiate treatment with a low-dose of CVN424 on Day 1; the low-dose arm will continue to receive their low dose each day, while the high-dose arm will increase their daily dosage to the high-dose CVN424 beginning on Day 8 ±2 days and continuing thereafter. Study drug will be self-administered each morning as an oral suspension. Subjects will continue their other PD medications.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult who is 30 to 80 years of age inclusive at study entry.
* Has idiopathic Parkinson's disease, Hoehn and Yahr stages 2-4, and is on a stable dosage of levodopa.
* Experiences an average of at least 2 h total OFF time/day, and at least 1 h each day, per Patient Motor Diary over 2 days during Screening assessment.
* The subject signs and dates a written informed consent form (ICF) and any required privacy authorization prior to the initiation of any study procedures.

Exclusion Criteria:

* Has atypical parkinsonism, severe disabling dyskinesia, or severe motor fluctuations that the investigator considers likely to interfere with study participation or assessments, or history of implant for Deep Brain Stimulation.
* Poor concordance (<75%) of self-report with site rater on in-clinic Screening period Patient Motor Diary. Subjects with low concordance may be retested after further instruction, at investigator's discretion.
* Screening period Patient Motor Diary scored at-home over 2 days demonstrates unacceptable quality of the diary, with more than 4 errors per day. (Assistance from caregivers is permitted if they also will be providing assistance with home Patient Motor Diary entries for Day 15 and 27 efficacy assessments.) Subjects with more than 4 errors per day may be retested after further instruction, at investigator's discretion.
* Body mass index (BMI) at Screening <18.0 or >35.0 kg/m2, inclusive.
* Subject has evidence of Clinically significant neurologic or other disorder or impairment that, in opinion of Investigator, is reasonably expected to impact the ability of the subject to participate or to confound the study results.
* Subject has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (i.e., a history of malabsorption, any surgical intervention known to impact absorption [e.g., bariatric surgery or bowel resection]).
* Subject has a history of cancer or other malignancy, with the exception of low-grade cervical intraepithelial neoplasia, low-grade (low-risk) prostate cancer, or 5-year cancer-free survivors of basal or squamous cell carcinoma, higher-grade cervical intraepithelial neoplasia or prostate cancer.
* Has a history of human immunodeficiency virus (HIV) infection.
* Subject has a supine blood pressure outside the ranges of 80 to 160 mm Hg for systolic and 50 to 100 mm Hg for diastolic, confirmed with up to two repeat tests, at the Screening Visit; or symptomatic orthostatic hypotension, in the opinion of the investigator.
* Subject has a resting heart rate outside the range 50 to 100 bpm, confirmed with up to two repeat tests, at the Screening Visit.
* Positive urine result for illegal drugs (except cannabis) at Screening, or history of illegal drug use (except cannabis) or alcohol abuse within 1 year prior to the Screening Visit.
* Subject has received any investigational compound (defined as a drug that has not been FDA-approved) within 30 days prior to the first dose of study medication, or within 5 half-lives of the investigational compound, whichever is greater.
* Subject has, within the prior month, ingested any excluded medication, supplements, or food products listed in the Excluded Medications and Dietary Products table as listed in Table 2.
* Male subjects who do not agree to all the following rules: when sexually active with female partner(s) of childbearing potential during the study and for 12 weeks after the last dose of study drug: a) use an acceptable method of birth control (condom with spermicide or surgical sterilization) and b) refrain from sexual activity with female partners who do not use an acceptable method of birth control. Barrier contraception (condom with spermicide) must be used by all male subjects who were not surgically sterilized at least 90 days prior to screening. Male subjects must also agree to refrain from sperm donation during the study and until 12 weeks after the last dose of study drug.
* Female subjects who are pregnant or breastfeeding or plan to become pregnant or donate ova during the study or for 30 days after the last dose of study drug. Women of childbearing potential (WOCBP) also must be practicing an adequate method of birth control (e.g., oral or parenteral contraceptives, intrauterine device, barrier, abstinence).
* Risk of suicide according to the investigator's clinical judgment or has made a suicide attempt in the previous 3 years.
* Subject is a study site employee or an immediate family member of a study site employee

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-11-06 (Actual); Study Completion 2021-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Kapurch, Study Chair — Cerevance, Inc.
Locations (21):
- United States (21):
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - SC3 Research - Pasadena, Pasadena, California
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Nova Clinical Research, Bradenton, Florida
  - Premier Clinical Research Institute, Miami, Florida
  - Parkinson's Disease Treatment Center of SW Florida, Port Charlotte, Florida
  - Accel Research Site - Brain and Spine Institute of Port Orange, Port Orange, Florida
  - USF Parkinson's Disease and Movement Disorders Center, Tampa, Florida
  - Charter Research, Winter Park, Florida
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - Parkinson's Disease and Movement Disorder Center, Kansas City, Kansas
  - Boston Clinical Trials, Roslindale, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - Bio Behavioral Health, Toms River, New Jersey
  - New York Neurology Associates, New York, New York
  - M3 Wake Research, Raleigh, North Carolina
  - Optimed Research Ltd, Columbus, Ohio
  - Neurology Diagnostics Inc, Dayton, Ohio
  - Prisma Health, Greenville, South Carolina
  - Central Texas Neurology Consultants, Round Rock, Texas
  - Inland Northwest Research, LLC, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 21 study sites in the United States
Groups:
- Placebo Arm: Participants were randomized in a 1:1:1 ratio into 1 of 3 study arms to receive either once daily (QD) low-dose CVN424 (50 milligrams [mg]), high-dose CVN424 (150 mg), or matching placebo.
- CVN424 50 mg; CVN424 150 mg: Participants were randomized in a 1:1:1 ratio into 1 of 3 study arms to receive either QD low-dose CVN424 (50 mg), high-dose CVN424 (150 mg), or matching placebo.
Period: Overall Study
Arm/Group | Placebo Arm | CVN424 50 mg | CVN424 150 mg
Started (Number of patients to be enrolled.) | 44 | 45 | 47
Completed | 41 | 42 | 44
Not Completed | 3 | 3 | 3
Not completed — Withdrawal by Subject | 2 | 2 | 1
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set comprised of all participants who were enrolled and received at least 1 dose of study drug, classified according to the treatment they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Arm | CVN424 50 mg | CVN424 150 mg | Total
Number analyzed (Participants) | 44 | 45 | 47 | 136
Age, Continuous [Median (Full Range); unit: years] | 67 [47 to 80] | 63 [46 to 78] | 65.6 [35 to 80] | 65.2 [35 to 80]
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (7.10) | 63.0 (7.67) | 65.6 (9.05) | 65.2 (8.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 20 | 42
  Male | 34 | 33 | 27 | 94
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 1 | 5
  White | 42 | 41 | 46 | 129
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) Related to Study Drug
Description: An adverse event is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. TEAEs are defined as any event with onset during or after the first dose of study treatment (active or placebo).
Time Frame: Up to Day 35
Population: Safety Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Arm | CVN424 50 mg | CVN424 150 mg
Number analyzed (Participants) | 44 | 45 | 47
Percentage of participants | 9.1 | 17.8 | 19.1

2. Secondary Outcome: Percentage of Participants With Clinically Significant Abnormal Laboratory Parameters
Description: Blood and urine samples were collected for the analysis of laboratory parameters including clinical chemistry, hematology, and urinalysis. The investigator was responsible for reviewing laboratory results for clinically significant abnormalities.
Time Frame: Up to Day 35
Population: Safety Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Arm | CVN424 50 mg | CVN424 150 mg
Number analyzed (Participants) | 44 | 45 | 47
Percentage of participants | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants With Clinically Significant Changes 12-Lead Electrocardiogram (ECG) Findings
Description: 12-lead ECG recordings including heart rate and measured PR, QRS, QT, QT interval with Fridericia's correction method (QTcF) and QT interval with Bazett's correction method (QTcB) intervals. 12-lead ECG recordings were obtained after participants rested for at least 5 minutes in supine position. The investigator was responsible for reviewing laboratory results for clinically significant abnormalities.
Time Frame: Up to Day 35
Population: Safety Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Arm | CVN424 50 mg | CVN424 150 mg
Number analyzed (Participants) | 44 | 45 | 47
Percentage of participants | 0 | 0 | 0

4. Secondary Outcome: Percentage of Participants With Clinically Significant Abnormal Vital Signs
Description: Vital signs including blood pressure (systolic and diastolic blood pressure), pulse rate, body temperature, respiratory rate and weight were measured after participants rested for at least 5 minutes in supine position. The investigator was responsible for reviewing laboratory results for clinically significant abnormalities.
Time Frame: Up to Day 35
Population: Safety Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Arm | CVN424 50 mg | CVN424 150 mg
Number analyzed (Participants) | 44 | 45 | 47
Percentage of participants | 0 | 0 | 0

5. Secondary Outcome: Change From Baseline in 2-day Average OFF Time
Description: The Patient Motor Diary data (Hauser Diary) was completed by the participant to record the broad motor symptoms of pharmacodynamics. Categories included time asleep, OFF time, ON time without dyskinesia, ON time with non-troublesome dyskinesia, and ON time with troublesome dyskinesia. These diaries were collected for 24 hours on each of 2 consecutive days with records for every 30 minutes interval. The average daily OFF time was calculated from the records with reported OFF time. Baseline was defined as Day 0. Change from Baseline was defined as post Baseline minus Baseline value.
Time Frame: Baseline and at Day 27
Population: Primary Efficacy Analysis Set comprised of all participants who were eligible, randomized, and received at least one dose of study drug, classified according to the treatment actually received. Only those participants with data available at specified timepoints has been presented.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Placebo Arm | CVN424 50 mg | CVN424 150 mg
Number analyzed (Participants) | 39 | 38 | 44
Hours | -0.462 (2.9265) | -1.342 (2.9680) | -1.563 (2.5261)

ADVERSE EVENTS:
Time Frame: Up to Day 35
Description: TEAEs has been collected in Safety Analysis Set.
Arm/Group | Placebo Arm | CVN424 50 mg | CVN424 150 mg
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/45 | 1/47
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/45 | 1/47
Other Adverse Events (participants affected / at risk) | 4/44 | 8/45 | 9/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Arm (N=44) | CVN424 50 mg (N=45) | CVN424 150 mg (N=47)
cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — The SAE unrelated to study treatment was an event of cardiac arrest in 1 (2.1%)patient in the CVN424 150 mg group that led to study drug discontinuation and death.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Arm (N=44) | CVN424 50 mg (N=45) | CVN424 150 mg (N=47)
Nausea (Gastrointestinal disorders) | 0 | 2 | 2
Headache (Nervous system disorders) | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0
Gamma-glutamyl transferase increased (Investigations) | 0 | 1 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Behaviour disorder (Psychiatric disorders) | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 1
Nightmare (Psychiatric disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT04191577/Prot_SAP_000.pdf